CLINICAL TRIAL: NCT01034410
Title: An Open-label Randomized Controlled Phase II Study of AS1411 Combined With Cytarabine in the Treatment of Patients With Primary Refractory or Relapsed Acute Myeloid Leukemia
Brief Title: A Study of AS1411 Combined With Cytarabine in the Treatment of Patients With Primary Refractory or Relapsed Acute Myeloid Leukemia
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Antisoma Research (Industry)
Responsible Party: Fredrik Erlandsson, MD, Antisoma
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: AS1411-C-203
Record Dates: First submitted 2009-12-16; First posted 2009-12-17 (Estimated); Last update posted 2011-02-02 (Estimated); Status verified 2011-02

CONDITIONS: Acute Myeloid Leukemia
Keywords: AS1411; AML; relapsed; refractory; aptamer; nucleolin
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Recurrence | interventions — AGRO 100; Cytarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control (Active Comparator): cytarabine 2g/m2 bid Days 4-7
  Interventions: Drug: Cytarabine
- AS1411-40 (Experimental): AS1411 40mg/kg/day d1-7 plus cytarabine 2g/m2 bid days 4-7
  Interventions: Drug: AS1411; Drug: Cytarabine
- AS1411-80 (Experimental): AS1411 80mg/kg/day d1-7, cytarabine 2g/m2 bid days 4- 7/ bid d4-7
  Interventions: Drug: AS1411; Drug: Cytarabine

INTERVENTIONS:
Drug: AS1411 — AS1411 40mg/kg/day or AS1411 80mg/kg/day
  Arms: AS1411-40; AS1411-80
Drug: Cytarabine — Cytarabine 2g/m2 bid Days 4-7
  Other Names: Ara-C

SUMMARY:
This is an open label randomized controlled phase II study of AS1411 combined with Cytarabine in the treatment of patients with primary refractory or relapsed acute myeloid leukemia.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of AML as defined by the World Health Organization (WHO) classification (Vardiman 2009)
* Primary refractory AML (defined as a failure to achieve a CR or CRi after therapy with curative intent) or AML in first relapse
* ECOG Performance status 0, 1 or 2
* Age > 18 and < 70 years
* For patients presenting with primary refractory AML, > 20% blasts on baseline bone marrow assessment
* For patients presenting with relapsed AML, > 5% blasts on baseline bone marrow assessment

Exclusion Criteria:

* An initial diagnosis of acute promyelocytic leukemia (as defined by French-American-British criteria (Bennett 1976))
* Secondary AML, defined as AML evolving from antecedent hematological disorder or prior exposure to leukemogenic therapy or agent
* Clinically active CNS leukemia
* Previously received a total cumulative dose of cytarabine > 6g/m2 in the last 6 months
* Previously received > 1 induction regimen (Defined as 1 or 2 cycles of a drug or a drug combination administered as remission induction therapy)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2010-01; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
To compare the response rate (CR + CRi) of AS1411 at 40 and 80mg/kg/day in combination with cytarabine therapy with the response rate (CR + CRi) of cytarabine therapy alone | Dec 2011

SECONDARY OUTCOMES:
To compare duration of remission, disease free survival and overall survival of AS1411 at 40 or 80mg/kg/day in combination with cytarabine therapy with that of cytarabine alone. | Dec 2011
To compare the time to hematological recovery of AS1411 at 40 or 80mg/kg/day in combination with cytarabine therapy with that of cytarabine alone. | Dec 2011
To compare the safety of AS1411 at 40 or 80mg/kg/day in combination with cytarabine therapy with that of cytarabine alone. | Dec 2011
To evaluate and compare a range of PD markers in patients administered AS1411 in combination with cytarabine therapy with the same PD markers in patients administered cytarabine therapy alone. | Dec 2011
To further define the PK of AS1411 | Dec 2011

CONTACTS AND LOCATIONS:
Overall Officials: Rob Stuart, MD, Principal Investigator — Medical University of South Carolina
Locations (14):
- United States (3):
  - UCLA, Los Angeles, California
  - Weill Medical College of Cornell University, New York, New York
  - Medical University of South Carolina, Charleston, South Carolina
- Australia (5):
  - Royal North Shore Hospital, St Leonards, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Royal Adelaide Hospital, Adelaide, South Australia
  - The Alfred Hospital, Melbourne, Victoria
  - Royal Perth Hospital, Perth, Western Australia
- Christchurch Hospital, Christchurch, New Zealand
- Taiwan (5):
  - Changhua Christian Hospial, Changhua, Changhua Country
  - China Medical University Hospital, Taichung
  - Taipei Veterans General Hospital, Taipei
  - Tri-Service General Hospital, Taipei
  - National Taiwan University Hospital, Taipei